CLINICAL TRIAL: NCT06922539
Title: A Phase 1a/1b Trial in Relapsed/Refractory Small Cell Lung Cancer to Determine the Safety Profile, Pharmacology, and Maximum Tolerated Dose of ST-001, a Fenretinide Phospholipid Suspension (12.5 mg/mL) for Intravenous Infusion
Brief Title: ST-001 nanoFenretinide in Relapsed/ Refractory Small Cell Lung Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: SciTech Development, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ST-001-020
Record Dates: First submitted 2025-03-22; First posted 2025-04-10 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Small Cell Lung Cancer
Keywords: fenretinide; SCLC; Relapsed/Refractory; Relapsed/Refractory SCLC; R/R SCLC; ST-001; intravenous administration
MeSH Terms: conditions — Small Cell Lung Carcinoma; Recurrence | interventions — Fenretinide; MAC-ST-001

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Standard Phase 1a (Experimental): During the Standard Phase 1a, three patients are enrolled into each dose level cohort and the three patients must be evaluated for cycle 1 toxicity before the decision can be made to open the next higher dose level.
  Interventions: Drug: Fenretinide
- Expanded Phase 1b (Experimental): Expansion of the dose-finding Phase 1a to determine the safety and maximum tolerated dose (MTD) of the investigative drug product (ST-001).
  Interventions: Drug: Fenretinide

INTERVENTIONS:
Drug: Fenretinide — Intravenous administration
  Other Names: ST-001
  Arms: Standard Phase 1a
Drug: Fenretinide — Intravenous administration
  Other Names: ST-001
  Arms: Expanded Phase 1b

SUMMARY:
This study evaluates a fenretinide phospholipid suspension for the treatment of small cell lung cancer (SCLC).

DETAILED DESCRIPTION:
Fenretinide has been shown to be a relatively safe and effective anticancer therapy; however, low fenretinide bioavailability and dose limiting toxicities due to excipients used in previous formulations has impeded its therapeutic utility. The product formulation in the current study (ST-001) is a phospholipid suspension of nanoparticle sized fenretinide. The current study is a Phase 1 trial in in relapsed/refractory small cell lung cancer to determine the safety profile, pharmacology, and maximum tolerated dose (MTD) of ST-001.

ELIGIBILITY:
Inclusion Criteria:

* Small cell lung cancer (SCLC).
* Patients must all have at least one measurable disease site using RECIST version 1.1 criteria.
* Patients must have had prior treatment with radiation therapy or with platinum-based chemotherapy ± immunotherapy with no limit on the number of prior systemic treatment regimens.
* Relapsed/refractory disease of any stage if incurable in nature, is eligible for enrollment.
* Minimum of 4 weeks must have elapsed since last systemic treatment or radiation therapy treatment (or 6 weeks for any nitrosourea-containing regimens), and patients must have recovered from all toxicity of last treatment and cleared the pharmacological agent(s) used previously.
* ECOG performance status 0-1 (Karnofsky ≥60%).
* Life expectancy greater than 6 months.
* Patients must have normal organ and marrow function.
* Triglyceride blood level (fasting) <300mg/dL at time of enrollment (normal: <150mg/dL; borderline high = 150-199mg/dL; high = 200-499mg/dL; very high = 500mg/dL or higher).
* Women of non-child bearing potential, that is women who have been menopausal or surgically sterile for more than 1 year, are eligible for enrolment in the study.
* Informed consent of the patient or a legal authorized representative (LAR) must be obtained prior to any study related procedures.

Exclusion Criteria:

* Mixed SCLC/NSCLC tumors are not eligible. Pregnant or breastfeeding women cannot take part in this study. Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier.
* Patients who are receiving any other investigational agents. SCLC patients with history of CNS metastasis may be included if CNS disease is asymptomatic and controlled without progression at least 4 weeks after treatment with radiotherapy, and patient is either no longer taking corticosteroids or on a stable dose of corticosteroids.
* History of allergic reactions or sensitivity to retinoids or to any excipients of ST-001.
* Patients who require concurrent treatment with drugs that are strong CYP3A inducers are excluded from the trial.
* Patients who require concurrent treatment with drugs that are strong to moderate CYP3A inhibitors are excluded from the trial.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure (NY heart classification III/IV), unstable angina pectoris, cardiac arrhythmia, QTc interval >450 milliseconds for men and >460 milliseconds for women on baseline triplicate ECG, or psychiatric illness/social situations that would limit compliance with study requirements.
* HIV-positive patients on combination antiretroviral therapy are ineligible. Patients with any active hepatitis infections. Presence of nyctalopia (night blindness), or hemeralopia (defective vision in a bright light, 'day blindness') at enrollment, or any other retinal, ophthalmological condition (e.g.: retinitis pigmentosa, choroidoretinitis and xerophthalmia), and glaucoma.
* History of solid tumor malignancy other than the diseases under study, diagnosed within the last three (3) years of study enrollment, excluding adequately treated basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer, in situ breast cancer, in situ prostate cancer (patients must have shown no evidence of active disease for 2 years prior to enrollment).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2025-12-11 (Actual); Primary Completion 2027-05-01 (Estimated); Study Completion 2028-10-01 (Estimated)

PRIMARY OUTCOMES:
To determine the MTD of ST-001 (12.5mg/mL) for IV infusion in patients with SCLC | From enrollment to end of treatment is 3 weeks
  To determine the maximum tolerated dose (MTD) and dose limiting toxicity (DLT) of ST-001 12.5 mg/mL for IV infusion (ST-001) in patients with Relapsed/Refractory SCLC when ST-001 is administered via 4-hour IV infusion daily for five consecutive days, q3weeks. MTD reflects the highest dose of drug that did not cause a Dose-Limiting Toxicity (DLT) in >33% of participants. DLTs are defined as any treatment-related Common Terminology Criteria for Adverse Events Version 5.0 (CTCAE 5.0) Grade 3 or 4 adverse events.

SECONDARY OUTCOMES:
To describe the toxicity profile of ST-001 in patients with SCLC | From enrollment to end of treatment is 3 weeks
  Determine the number of participants with treatment-related adverse events as assessed by CTCAE v5.0
To observe and record anti-tumor activity of ST-001 in patients with SCLC | From enrollment to end of treatment is 3 weeks
  Preclinical studies with fenretinide suggest potential efficacy against SCLC. Patients will be carefully monitored for tumor response and symptom relief in addition to safety and tolerability. Objective Response Rate (ORR) and progression-free survival (PFS) will be used as tumor response endpoints in this study.
Objective Response Rate (ORR) | From enrollment to end of treatment is 3 weeks
  ORR = (Number of patients with complete or partial response) / (Total number of evaluable patients) x 100. Minimum duration of individual patient participation is 3 weeks (one cycle of therapy) to be evaluable for response.
Progression-free survival (PFS) | From enrollment to end of treatment is 3 weeks
  PFS is defined as the time from start of treatment to disease progression (increase in tumor size, new metastases) or death.
To describe the pharmacokinetics of fenretinide when ST-001 is administered by daily infusion for 5 consecutive days every 3 weeks. | From enrollment to end of treatment is 3 weeks
  The endpoint for the pharmacokinetic studies is to assess fenretinide blood plasma levels as a function of administered dose and to determine the following PK parameters: maximum fenretinide concentration (Cmax), time of Cmax (Tmax), volume of distribution (Vd), clearance (CL), elimination and fenretinide half-life (t½).
Cmax | From enrollment to end of treatment is 3 weeks
  Peak plasma fenretinide concentration (in ng/mL)
Tmax | From enrollment to end of treatment is 3 weeks
  The time it takes for fenretinide to reach the maximum concentration (Cmax) after drug administration (in hours)
Vd | From enrollment to end of treatment is 3 weeks
  Volume of distribution; fenretinide's propensity to either remain in the plasma or redistribute to other tissue compartments (in liters)
t½ | From enrollment to end of treatment is 3 weeks
  Fenretinide elimination and half-life; the time it takes for the amount of a drug's active substance in your body to reduce by half (hours)

CONTACTS AND LOCATIONS:
Overall Officials: Ali Moiin, MD, Study Director — SciTech Development, Inc.
Locations (1):
- University of Southern California, Los Angles, California, United States

IPD SHARING:
Plan to Share IPD: No